CLINICAL TRIAL: NCT06224036
Title: A Randomized, Open, Multicenter, Phase IIa Clinical Study on the Early Bactericidal Activity, Safety, Tolerance and Pharmacokinetics of JDB0131 Benzenesulfonate Tablets in Drug Sensitive Pulmonary Tuberculosis Patients
Brief Title: Clinical Study of JDB0131 Benzenesulfonate Tablets in Patients With Drug-sensitive Pulmonary Tuberculosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chest Hospital (Other)
Collaborators: West China Hospital (Other); Wuhan Pulmonary Hospital (Other)
Responsible Party: Principal Investigator, Chu naihui, TB Director, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JDB-131-201
Record Dates: First submitted 2023-07-09; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Drug-resistant Tuberculosis
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — OPC-67683

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- First group (Experimental): JDB0131 Benzenesulfonate tablets,100mg BID group,12 cases
  Interventions: Drug: JDB0131
- Second group (Experimental): JDB0131 Benzenesulfonate tablets 200mg QD group,12 cases
  Interventions: Drug: JDB0131
- Third group (Experimental): JDB0131 Benzenesulfonate tablets 200mg BID group,12 cases
  Interventions: Drug: JDB0131
- Forth group (Active Comparator): Ethylpyrazine rifampicide (II) QD group,8 cases
  Interventions: Drug: Ethylpyrazine rifampicide (II)
- Fifth group (Active Comparator): Delamanid Tablets 100mg BID group,8 cases
  Interventions: Drug: Delamanid

INTERVENTIONS:
Drug: JDB0131 — JDB0131 benzenesulfonate is a new anti tuberculosis compound based on delamanid. According to the existing results of pre clinical in vitro activity, in vivo efficacy, pharmacokinetics and safety in human body, JDB0131 benzenesulfonate has the same in vivo efficacy, better lung tissue distribution and better safety as delamanid.
  In December 2016, JDB0131 obtained the drug clinical approval issued by the CFDA, and were approved the clinical stage research that development of drug-resistant tuberculosis adaptation.
  Arms: First group; Second group; Third group
Drug: Delamanid — Delamanid is a new drug developed by Otsuka Pharmaceutical Co., Ltd. in Japan to treat multidrug resistant tuberculosis. In 2014, Delamanid was conditionally approved for marketing by the European Medicines Agency and recommended for use in adult MDR-TB patients who cannot form an effective regimen due to drug resistance or tolerance reasons. In the same year, WHO recommended that Delamanid be conditionally used for long-term treatment of adult MDR-TB. In 2016, the WHO recommended widening the age range for Delamanid to 6-17 years old. In March 2018, Delamanid was listed in China.
  Arms: Fifth group
Drug: Ethylpyrazine rifampicide (II) — Ethylpyrazine rifampicide (II) is suitable for the first two months of intensive treatment of pulmonary tuberculosis with short-term therapy. This product is a compound preparation, consisting of 0.15g of rifampicin (C43H58N4O12), 0.075g of isoniazid (C6H7N3O), 0.4g of pyrazinamide (C5H5N3O), and 0.275g of ethambutol hydrochloride (C10H24N2O2 · 2HCl) per tablet.
  Arms: Forth group

SUMMARY:
A randomized, open, drug controlled design of experiments was used to evaluate the early bactericidal activity, safety, tolerance and pharmacokinetic characteristics of JDB0131 benzenesulfonate tablet taken orally by drug sensitive pulmonary tuberculosis patients. Five groups are proposed to be set up in this test (JDB0131 benzenesulfonate 100mg BID, JDB0131 benzenesulfonate 200mg QD, JDB0131 benzenesulfonate 200mg BID, anti tuberculosis drug fixed dose composite dosage QD is determined according to the weight of the study participants, and delamanid 100mg BID)

ELIGIBILITY:
Inclusion Criteria:

* (Those who must meet all the selection criteria can enter the group)

  1. Age of study participants: 18 years old≤ age ≤ 65 years old, male or female;
  2. Study participant weight: 40kg≤ body weight≤90kg
  3. Patients with clinically confirmed pulmonary tuberculosis, and have not received anti-tuberculosis therapy within 2 years, at least one positive sputum acid-fast bacilli smear (AFB at least 1+);
  4. Be willing to provide a blood sample for HIV testing;
  5. Non-lactating and non-pregnant women who agree to use highly effective contraception throughout the study period, and male study participants must agree to use appropriate contraceptive methods throughout the study period;
  6. The study participants fully understand the purpose, nature, methods and possible adverse reactions of the trial, voluntarily act as research participants, and sign informed consent;
  7. Those who are willing to complete the test according to the requirements of the program.

Exclusion Criteria:

* (Meet any of the following criteria will be excluded)

  1. Rifampicin resistance;
  2. Positive for human immunodeficiency virus (HIV) antibodies; positive for hepatitis B surface antigen (HBsAg); positive for hepatitis C virus (HCV) antibodies; positive for treponemal antibodies;
  3. Clear hepatobiliary disease, including but not limited to chronic active hepatitis and/or severe hepatic insufficiency; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the upper limit of normal; Total serum bilirub (TBIL) > 2 times the upper limit of normal;
  4. Have a history of kidney disease or manifestations related to renal disease: 1) history of unstable or rapidly progressive kidney disease; 2) Moderate/severe renal impairment or end-stage renal disease (eGFR<60mL/min/1.73m2); 3) Serum creatinine (Cr) ≥ 133 μmol/L (1.5 mg/mL) in men, Cr ≥ 124 μmol/L (1.4 mg/mL) in women;
  5. Have a family history of QT prolongation syndrome or are taking drugs that cause QT interval prolongation, such as: quinidine, procainamide, amiodarone, sotalol, etc.;
  6. ECG showed the following abnormalities: 1) QTcF>450 ms (corrected by Fridericia formula); 2) pathological Q wave (defined as >40ms or depth >0.4-0.5mV); 3) ECG suggests pre-excitation syndrome; 4) ECG suggests left bundle branch block or right bundle branch block; 5) ECG shows second- or third-degree heart block; 6) QRS duration > 120ms indoor conduction delay; 7) Sinus heart rate < bradycardia of 50bpm;
  7. Those who have any of the following cardiovascular diseases or other conditions within 6 months before enrollment: 1) myocardial infarction; 2) Cardiac surgery or coronary revascularization (coronary artery bypass grafting/percutaneous transluminal coronary angioplasty); 3) unstable angina; 4) congestive heart failure (New York Cardiology Society Cardiac Function Class III or IV); 5) transient ischemic attack or severe cerebrovascular disease;
  8. Anyone who is unable to comply with the uniform diet due to allergies or special dietary requirements;
  9. Those with a history of gastrointestinal surgery or resection that may affect the absorption and/or excretion of oral medications;
  10. Those who have abnormal ophthalmic examination during the screening period and are judged by the investigator to be unsuitable for participating in this trial;
  11. Depression: those with a score higher than 7 on the Hamilton Depression Scale (17 items, see Appendix 2);
  12. Those who are judged to have any unstable or severe cardiovascular, renal, liver, hematology, tumor, endocrine metabolism, psychiatric or rheumatic diseases and therefore consider them unsuitable to participate in this trial;
  13. Those who cannot control the consumption of alcohol or alcohol-containing products from 48 h before administration to the completion of the last pharmacokinetic blood sample collection, and do not consume any food or beverage containing or metabolizing caffeine or xanthines (such as coffee, strong tea, cola, chocolate);
  14. Patients who have used other clinical trial study drugs within 3 months prior to administration;
  15. Patients with a history of alcohol dependence or substance abuse within 6 months prior to screening, which the investigator believes may affect the safety of study participants and affect trial adherence;
  16. Use of psychotropic drugs such as barbiturates, opioids, and phenothiazines within 30 days;
  17. Chronic systemic corticosteroid therapy, defined as any dose of systemic corticosteroid therapy, cumulative use for more than 4 weeks in the 3 months prior to enrollment;
  18. Those who are allergic to any investigational drug or related substances confirmed by the clinical judgment of the investigator;
  19. Strong inducers or inhibitors of cytochrome P450 enzyme (e.g., carbamazepine, phenytoin, rifampicin, clarithromycin, ritonavir, ketoconazole, itraconazole, etc.) within 30 days before treatment;
  20. Women with a positive pregnancy test or breastfeeding during screening;
  21. Those who received live attenuated vaccine within 4 weeks before the study drug (except inactivated influenza vaccine such as seasonal influenza vaccine for injection);
  22. Any condition that, in the judgment of the investigator, affects the study participant's adherence to the study protocol, or incorporates any serious medical or psychological condition that may affect the interpretation of efficacy and safety data, or that the study participant's participation in the trial may affect his or her own safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
EBA | he change of TB bacterium burden in sputum from Day 0 to Day 2 and/or Day 14
  Early bactericidal activity (EBA), counted by daily log (CFU) change

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | average of 6 month
  An AE was defined as any new medical problem, or exacerbation of an existing problem, experienced by a participant while enrolled in the trial, whether or not it was considered drug-related by the investigator.
Percentage of Participants With Immediately Reportable Events (IREs) | average of 6 month
  An AE was considered serious if it was fatal; life-threatening; persistently or significantly disabling or incapacitating; required in-participant hospitalization or prolonged hospitalization; a congenital anomaly/birth defect; or other medically significant event that, based upon appropriate medical judgment, may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the outcomes listed above. The following were considered as IREs- serious adverse events (SAEs), pregnancies in trial participants or their partners, and all events involving overdose, misuse and abuse.problem, experienced by a participant while enrolled in the trial, whether or not it was considered drug-related by the investigator.
ECG | an average of 6 month
  ECG QT Interval
Safe tolerance | through study completion, an average of 6 month
  laboratory tests
Safe tolerance | through study completion, an average of 6 month
  Eye examination and depression scale scores
Tmax | Day 0 to Day 21
  Time to Reach Maximal Peak Plasma Concentration for JDB0131
Cmax | Day 0 to Day 21
  Maximal Peak Plasma Concentration for JDB0131
AUC0-24h | Day 0 to Day 21
  Area under plasma concentration time curve from initial administration to 12 hours for JDB0131
T Tss,max | Day 0 to Day 21
  Steady state peak time for JDB0131
Css,max | Day 0 to Day 21
  Steady state peak concentration for JDB0131
Css,min | Day 0 to Day 21
  Steady-state valley concentration for JDB0131
Css,avg | Day 0 to Day 21
  Mean steady-state blood drug concentration for JDB0131
t1/2,ss | Day 0 to Day 21
  Elimination half life for JDB0131
AUC0-12,ss | Day 0 to Day 21
  Area under the plasma concentration time curve from the last administration to 12 hours for JDB0131
AUC0-t,ss | Day 0 to Day 21
  Area under the plasma concentration-time curve from the last dose to the last measurable concentration time "t" for JDB0131
AUC0-∞,ss | Day 0 to Day 21
  Area under the plasma concentration-time curve from the last dose extrapolated to infinity for JDB0131
Vd,ss | Day 0 to Day 21
  Apparent volume of distribution for JDB0131
CL,ss | Day 0 to Day 21
  Oral clearance for JDB0131
Rac（Cmax） | Day 0 to Day 21
  Ratio of Cmax,ss at day 14 to Cmax at day 1
Rac（AUC） | Day 0 to Day 21
  AUC0-12,ss at day 14 compared to AUC0-12 at day 1
Fluctuation coefficient | Day 0 to Day 21
  Percent fluctuation at steady state = 100 * (Css, max - Css, min) / Css, avg.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Wuhan Chest Hospital (Wuhan Institute For Tuberculosis Control), Wuhan, Hubei
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No